CLINICAL TRIAL: NCT00461318
Title: Enhancing the Quality of Life and Independence of Persons Disabled by Severe Mental Illness Through Supported Employment
Brief Title: The Effectiveness of Supported Employment for People With Severe Mental Illness: an RCT in Six European Countries
Acronym: EQOLISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLRT-2001-00683
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Psychosis
Keywords: vocational rehabilitation; psychosis; cross country comparison
MeSH Terms: conditions — Psychotic Disorders | interventions — Palliative Care; Rehabilitation, Vocational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Individual placement and support (vocational rehabilitation)

SUMMARY:
The primary aim of the study was to determine the effectiveness of a form of supported employment, Individual Placement and Support (IPS) compared to existing good quality rehabilitation and vocational services for people with psychotic illnesses in terms of 'open' employment outcomes (in the competitive labour market), and to examine its relative effectiveness in the context of different European welfare systems and labour markets. The primary hypothesis was that IPS patients would be more likely to obtain open employment than control service patients. Secondary hypotheses were that they would be in open employment for longer than the control patients, and that they would not spend more time in hospital.

DETAILED DESCRIPTION:
An RCT was conducted in six European centres: London (UK), Ulm-Guenzburg (Germany), Rimini (Italy), Zurich (Switzerland), Groningen (the Netherlands) and Sofia (Bulgaria). Patients were included if they had a diagnosis of SMI (psychotic illness including bipolar disorder), were aged 18 to retirement age, had been ill and had major role dysfunction for at least two years, were living in the community at baseline, had not been in competitive employment in the preceding year and expressed the desire to enter competitive employment. They were randomly allocated to receive either IPS or the 'Vocational Service' (control service). Given the need to consider the impact of gender and work history on vocational outcomes (20), service allocation was stratified by centre, gender and work history (more or less than a month's competitive employment in the five years prior to baseline). Randomisation was conducted centrally using MINIM Version 1.5. A researcher at each centre recruited the patients, submitted them to the statistician for randomisation and received the allocation by email. The allocation sequence was concealed until the services had been assigned, but it was not possible for patients, professionals or researchers to be blind to service allocation thereafter.

ELIGIBILITY:
Inclusion Criteria:

* pscychotic illness of at least a years duration
* unemployed for at least a year

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300
Dates: Start 2003-04; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
sucessful employment for one day in the open labour market

SECONDARY OUTCOMES:
duration of employment
psychiatric hospitalisation
well-being

CONTACTS AND LOCATIONS:
Overall Officials: jocelyn catty, DPhil, Study Director — St Georges Medical School, university of london
Locations (1):
- Division of mental health, St Georges medical school, university of london, London, United Kingdom

REFERENCES:
- [Derived] Burns T, Catty J, Becker T, Drake RE, Fioritti A, Knapp M, Lauber C, Rossler W, Tomov T, van Busschbach J, White S, Wiersma D; EQOLISE Group. The effectiveness of supported employment for people with severe mental illness: a randomised controlled trial. Lancet. 2007 Sep 29;370(9593):1146-52. doi: 10.1016/S0140-6736(07)61516-5. PMID 17905167